CLINICAL TRIAL: NCT04131595
Title: Phase 1 Vaccination Trial to Evaluate Safety, Tolerability and Immunogenicity of a Recombinant MVA-BN-WEV Vaccine in Healthy Adult Subjects
Brief Title: Vaccination Trial of a Recombinant MVA-BN-WEV Vaccine in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: JPM CBRN Medical (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WEV-MVA-001
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Equine Encephalitis
MeSH Terms: conditions — Encephalomyelitis, Equine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MVA-BN-WEV Dose 1 (Experimental): Subjects in treatment Group 1 will receive 2 administrations 4 weeks apart with MVA-BN-WEV vaccine of 1 x 107 Inf.U in 0.5 mL.
  Interventions: Biological: MVA-BN-WEV Dose 1
- MVA-BN-WEV Dose 2 (Experimental): Subjects in treatment Group 2 will receive 2 administrations 4 weeks apart with MVA-BN-WEV vaccine of 1 x 108 Inf.U in 0.5 mL
  Interventions: Biological: MVA-BN-WEV Dose 2
- MVA-BN-WEV Dose 3 (Experimental): Subjects in treatment Group 3 will receive 2 administrations 4 weeks apart with MVA-BN-WEV vaccine of 2 x 108 Inf.U in 2 x 0.5 mL
  Interventions: Biological: MVA-BN-WEV Dose 3

INTERVENTIONS:
Biological: MVA-BN-WEV Dose 1 — 1 x 10^7 Inf.U MVA-BN-WEV vaccine
  Arms: MVA-BN-WEV Dose 1
Biological: MVA-BN-WEV Dose 2 — 1 x 10^8 Inf.U MVA-BN-WEV vaccine
  Arms: MVA-BN-WEV Dose 2
Biological: MVA-BN-WEV Dose 3 — 2 x 10^8 Inf.U MVA-BN-WEV vaccine.
  Arms: MVA-BN-WEV Dose 3

SUMMARY:
To assess safety and tolerability as well as immune responses to the MVA-BN-WEV vaccine in the 3 treatment groups receiving different doses.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male and female subjects ≥18 and ≤50 years of age at screening (SCR).
* 2. General good health, without clinically relevant medical illness, physical exam findings, or laboratory abnormalities, as determined by the investigator.
* 3. Prior to performance of any trial specific procedures, the subject has read, signed and dated an informed consent form (ICF), having been advised of the risks and benefits of the trial in a language understood by the subject, and has signed the Health Insurance Portability and Accountability Act authorization form (HIPAA).
* 4. Body mass index (BMI) ≥18.5 and ≤35.
* 5. Female subjects of childbearing potential and male subjects who are sexually active with a female partner of childbearing potential must agree to the use of an effective method of birth control from at least 30 days prior to administration of the vaccine to until 30 days after the last vaccination. A woman is considered of childbearing potential unless post-menopausal (defined as ≥12 months without a menstrual period at SCR) or surgically sterilize (bilateral oophorectomy, bilateral tubal ligation, hysterectomy). Acceptable contraception methods are restricted to abstinence (abstinence only acceptable if refraining from heterosexual intercourse during the entire period of 30 days prior to administration of the vaccine until 30 days after the last vaccination), double barrier contraceptives, vasectomy, intrauterine contraceptive devices or licensed hormonal products.
* 6. Women of Childbearing Potential (WOCBP) must have a negative serum pregnancy test at SCR.
* 7. Negative human immunodeficiency virus antibody test (anti-HIV), negative hepatitis B surface antigen (HBsAG) and negative antibody to hepatitis C virus.
* 8. Troponin I within normal limits at SCR.

Exclusion Criteria:

* 1. Pregnant or breast-feeding women.
* 2. Subject has an acute or chronic medical condition that, in the opinion of the investigator, would render the trial procedures unsafe or would interfere with the evaluation of the responses, including but not limited to, neurologic, cardiovascular, respiratory, hepatic, hematologic, rheumatologic, endocrine, gastrointestinal, renal, autoimmune, or immunosuppressive conditions.
* 3. Laboratory parameters (such as complete blood count, serum biochemistry including aspartate aminotransferase (AST), alanine amino transferase (ALT), alkaline phosphokinase (AP), bilirubin, or creatinine values), pulse rate and/or blood pressure, or electrocardiogram (ECG) outside normal range at SCR and deemed clinically relevant by the investigator.
* 4. History of or active autoimmune disease; persons with vitiligo or thyroid disease taking thyroid replacement are not excluded. History of Guillain-Barré syndrome or Reye's syndrome.
* 5. Known or suspected impairment of immunologic functions including, but not limited to, clinically significant liver disease, diabetes mellitus type I, moderate to severe kidney impairment. A known immunodeficiency syndrome.
* 6. Known or suspected previous smallpox vaccination or vaccination with a poxvirus-based vaccine.
* 7. Known or suspected previous alphavirus infections (Eastern Equine Encephalitis Virus (EEEV), Venezuelan Equine Encephalitis Virus (VEEV), Western Equine Encephalitis Virus (WEEV), Chikungunya).
* 8. History of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision at least 6 months prior to SCR that is considered to have achieved cure. Subjects with history of skin cancer must not be vaccinated at the previous tumor site.
* 9. Clinically significant mental disorder not adequately controlled by medical treatment.
* 10. Active or recent history of chronic alcohol abuse and/or intravenous and/or nasal drug abuse (within the time period of 6 months before SCR).
* 11. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. tris(hydroxymethyl)-amino methane, chicken embryo fibroblast proteins, gentamicin, ciprofloxacin.
* 12. Known allergy to eggs.
* 13. History of anaphylaxis or severe allergic reaction to any vaccine.
* 14. Having received any vaccinations or planned vaccinations with a live vaccine within 30 days prior to first or after last trial vaccination.
* 15. Having received any vaccinations or planned vaccinations with an inactivated vaccine within 14 days prior to first or after last trial vaccination.
* 16. Recent blood donation (including platelets, plasma and red blood cells) within 4 weeks prior screening, or planned blood donations during active trial phase (until EAP Visit).
* 17. Chronic systemic administration (defined as more than 14 days) of >5 mg prednisone (or equivalent)/day or any other immunemodifying drugs during a period starting 3 months prior to administration of the vaccine and ending at the last visit of the active treatment phase. The use of topical, inhaled, ophthalmic and nasal glucocorticoids is allowed.
* 18. Post organ transplant subjects whether or not receiving chronic immunosuppressive therapy.
* 19. Administration or planned administration of immunoglobulins and/or any blood products during a period starting 3 months prior to administration of the vaccine and ending at the last visit of the active treatment phase. Receipt of packed red blood cells given for an emergent indication in an otherwise healthy person, and not required as ongoing treatment is not exclusionary (for example packed red blood cells emergently given during an elective surgery).
* 20. History of coronary heart disease, myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, significant arrhythmia with or without corrective/ablative surgery, or any other heart condition under the care of a doctor.
* 21. Use of any investigational or non-registered drug or vaccine other than the trial vaccine within 30 days preceding the first dose of the trial vaccine, or planned administration of such a drug during the trial period until the Follow-Up (FU) Visit 6 months after the last vaccination visit.
* 22. Clinical trial site personnel involved in this trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: Number of subjects reporting any serious adverse events (SAE) | within 7 months after vaccinations of subjects
  Number of subjects reporting any serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Fierro, MD, Principal Investigator — JCCT
Locations (1):
- Johnson County Clin-Trials, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fierro C, Weidenthaler H, Vidojkovic S, Schmidt D, Gafoor Z, Stroukova D, Zwiers S, Muller J, Volkmann A. Safety and immunogenicity of a novel trivalent recombinant MVA-based equine encephalitis virus vaccine: A Phase 1 clinical trial. Vaccine. 2024 Apr 11;42(10):2695-2706. doi: 10.1016/j.vaccine.2024.03.011. Epub 2024 Mar 16. PMID 38494412